CLINICAL TRIAL: NCT01715909
Title: An Open-Label, Randomized, Adaptive, Two-Arm, Multicenter Trial to Evaluate Pharmacokinetics And Pharmacodynamics of Two Doses of Oseltamivir (Tamiflu®) in The Treatment Of Influenza in Immunocompromised Children Less Than 13 Years Of Age, With Confirmed Influenza Infection
Brief Title: A Pharmacokinetic/Pharmacodynamic Study of Oseltamivir in Immunocompromised Children With Confirmed Influenza Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NV25719; 2012-002633-11 (EudraCT Number)
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

ARMS (2):
- Oseltamivir: Standard dose (Experimental): Participants will receive standard dose of oseltamivir capsules or suspension orally for 5 to maximum of 20 days depending on weight. Infants <1 year of age will receive oseltamivir at a dose of 3 milligrams per kilogram (mg/kg).
  Interventions: Drug: Oseltamivir
- Oseltamivir: Triple dose (Experimental): Participants will receive three times the standard dose of oseltamivir capsules or suspension orally for 5 to maximum of 20 days depending on weight and age. Infants <1 year will receive standard dose at 3 mg/kg.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Participants will receive standard dose (30 to 75 milligrams [mg]) or triple standard dose (90 to 225 mg) of oseltamivir orally daily for up to maximum of 20 days. Standard dose of oseltamivir according to weight (except infants): 30 mg twice daily for </= 15 kilograms (kg) body weight participants; 45 mg twice daily for 15 to 23 kg body weight participants; 60 mg twice daily for 23 to 40 kg body weight participants; and 75 mg twice daily for greater than (>) 40 kg body weight participants. Standard dose for infants is 3 mg/kg.
  Other Names: Tamiflu

SUMMARY:
This open-label, randomized, adaptive, 2-arm, multicenter study will evaluate the pharmacokinetics and pharmacodynamics of oseltamivir (Tamiflu) in immunocompromised children, less than (<) 13 years of age, with confirmed influenza infection. Participants will be randomized to receive either the standard dose or triple dose of oseltamivir orally daily for a minimum of 5 days and up to 20 days. Infants <1 year of age will be randomized to the standard dose arm only.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children, <13 years of age
* Rapid influenza diagnostic test (RIDT), polymerase chain reaction (PCR), or viral culture positive for influenza
* Immunocompromised
* Symptoms/signs suggestive of influenza like illness (ILI)
* Less than or equal to (</=) 96 hours between onset of ILI and first dose of study drug

Exclusion Criteria:

* Clinical evidence of severe hepatic impairment
* Infants with post-menstrual age (PMA) <36 weeks
* Clinical evidence of significant renal impairment
* Allergy to oseltamivir or excipients
* Hereditary fructose intolerance
* Received anti-viral treatment with activity against influenza (for example amantadine, rimantadine, oseltamivir, laninamivir, peramivir, zanamivir, and ribavirin) or probenecid medication within 2 weeks prior to randomization

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2014-01-22 (Actual); Primary Completion 2018-06-17 (Actual); Study Completion 2018-06-17 (Actual)

PRIMARY OUTCOMES:
Steady State Area Under the Concentration-Time Curve From Time 0 to 12 Hours (AUC0-12) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Steady State AUC0-12 of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Maximum Plasma Concentration (Cmax) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Cmax of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Trough Plasma Concentration (Ctrough) of Oseltamivir | Pre-dose (within 30 minutes prior to administration) on Days 3 or 4
Ctrough of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration) on Days 3 or 4
Time to Cessation of Viral Shedding, as Assessed by Polymerase Chain Reaction (PCR) or Culture Testing | From randomization to negative PCR/culture test result (up to Day 50)

SECONDARY OUTCOMES:
Time to Resolution of Influenza Symptoms (including fever),, as Assessed by Canadian Acute Respiratory Infections Scale (CARIFS) | From randomization to resolution of all influenza symptoms (up to Day 50)
Number of Participants With Adverse Events | Baseline up to Day 50
Number of Participants With Influenza Associated Complications | Baseline up to Day 50
Number of Participants With Viral Resistance | Baseline up to Day 50
Half-life (t1/2) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
t1/2 of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Time to Maximum Concentration (Tmax) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Tmax of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Elimination Rate Constant (Ke) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Ke of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Apparent Volume of Distribution (V/F) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
V/F of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Apparent Clearance (CL/F) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
CL/F of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Time to Last Measurable Concentration (Tlast) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Tlast of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Last Measurable Concentration (Clast) of Oseltamivir | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4
Clast of Oseltamivir Carboxylate | Pre-dose (within 30 minutes prior to administration), 1.5, 4, 8 hours post-dose on Days 3 or 4

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (50):
- United States (7):
  - Lucile Packard Child Hosp; Pediatric Pulmonary Division, Palo Alto, California
  - The Children's Hospital; Pediatric Infectious Diseases, Aurora, Colorado
  - Tufts Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Seattle Children's Hospital, Seattle, Washington
- Belgium (3):
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (4):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Graacc-Grupo de Apoio ao adolescente e a crianca com cancer, São Paulo, São Paulo
  - Casa de Saúde Santa Marcelina, São Paulo, São Paulo
- Canada (3):
  - Children'S Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital For Sick Children; Infectious Disease Dept, Toronto, Ontario
  - McGill University; Montreal Children's Hospital; Oncology, Montreal, Quebec
- Hospital Dr. Gustavo Fricke, Viña del Mar, Chile
- Colombia (2):
  - Centro Medico Imbanaco, Cali
  - Fundacion Clinica Valle de Lili, Department Rheumatology, Cali
- Turun yliopistollinen keskussairaala, Turku, Finland
- Germany (5):
  - Charité - Universitätsmedizin Berlin;Klinik für Allgemeine Pädiatrie, Berlin
  - Universitatsklinikum Frankfurt, Frankfurt
  - Dr. Von Haunersches Kinderspital, München
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen UNI-Klinik für Kinder- und Jugendmedizin, Tübingen
- Greece (2):
  - Childrens Regional Hospital Aglaia Kyriakou, Athens
  - Aghia Sophia Children's Hospital; Pediatric Rheumatology Unit; 1st Department of Pediatrics, Athens
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Schneider Children's Medical Center of Israel; Pediatrics Department, Petah Tikva
  - The Chaim Sheba Medical Center; Multiple Sclerosis Center, Ramat Gan
  - The Dana Children's Hospital, Tel Aviv
- Italy (3):
  - Ospedale Pediatrico Bambino Gesu, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico; Unità Operativa Complessa Pediatria 1, Milan, Lombardy
  - ASST DI MONZA; Divisione Malattie Infettive, Monza, Lombardy
- Mexico (2):
  - Instituto Nacional de Pediatria; Departmento de Neurologia, México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez; Universidad Autónoma de Nuevo León, Monterrey
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Children Hospital, Olsztyn; Ward of Pediatric Hematology and Oncology, Olsztyn
  - Samodzielny Publiczny Szpital Kliniczny nr 1 im. prof.Tadeusza Sokolowskiego, Szczecin
  - Medical University of Silesia; Department of Pediatric Hematology and Oncology, Zabrze
- South Africa (3):
  - Tygerberg Hospital; Rheumatology, Cape Town
  - WWCT Lakeview Hospital, Johannesburg
  - Chris Hani Baragwanath Hospital, Johannesburg
- Spain (5):
  - Hospital Sant Joan De Deu, Esplugues de Llobregas, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario La Paz, Madrid